CLINICAL TRIAL: NCT05674461
Title: The Effect of WhatsApp-based and Face-to-Face Education and Counseling on Women's Quality of Life and Traditional Practices in the Postpartum Period
Brief Title: The Effect of Education and Counseling on Women's Quality of Life and Traditional Practices in the Postpartum Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gamze DERMAN, PhD student, Inonu University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20224107
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Postpartum Period
Keywords: Quality of life; Traditional practice; Training; WhatsApp; Face-to-face
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WhatsApp Group (Experimental): In the study, training modules including general information about the postpartum period, breastfeeding counseling, postpartum nutrition, puerperal psychology, family planning and postpartum exercises, consisting of 4 sessions, will be applied to the women in the experimental group.
  Trainings will be sent to the women in the WhatsApp experimental group in the form of videos via the WhatsApp application. The videos will be prepared with the researchers' own voice and image. Each training video will be sent for 15-30 minutes (in the form of short videos, if necessary, divided into parts).
  Women will be supported through messages in order to increase their motivation and provide counseling regarding their possible questions and problems.
  Interventions: Other: WhatsApp Group
- Face-to-face Group (Experimental): In the study, training modules including general information about the postpartum period, breastfeeding counseling, postpartum nutrition, puerperal psychology, family planning and postpartum exercises, consisting of 4 sessions, will be applied to the women in the experimental group.
  The trainings will be given to the women in the experimental group face-to-face by the researchers in the form of 15-30 minute trainings in their own home environment.
  Women will be supported through messages in order to increase their motivation and provide counseling regarding their possible questions and problems.
  Interventions: Other: Face-to-face Group
- Control (Other): No intervention will be applied to the mothers in the control group.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: WhatsApp Group — Each of the women will be informed about the purpose and content of the study at the first meeting, and informed consent will be obtained from the women who meet the conditions for participation and agree to participate. The pre-test data in the research will be obtained with the Participant Identification Form and WHOQOL-BREF-TR Trainings will be sent to the women in the WhatsApp experimental group in the form of videos via the WhatsApp application. The videos will be prepared with the researchers' own voice and image. Each training video will be sent for 15-30 minutes (in the form of short videos, if necessary, divided into parts). At the end of the 2nd and 6th months, the final test data will be obtained by completing the Participant Identification Form and WHOQOL-BREF-TR
  Arms: WhatsApp Group
Other: Face-to-face Group — Each of the women will be informed about the purpose and content of the study at the first meeting, and informed consent will be obtained from the women who meet the conditions for participation and agree to participate. The pre-test data in the research will be obtained with the Participant Identification Form and WHOQOL-BREF-TR The trainings will be given to the women in the experimental group face-to-face by the researchers in the form of 15-30 minutes of training in their own home environment. At the end of the 2nd and 6th months, the final test data will be obtained by completing the Participant Identification Form and WHOQOL-BREF-TR
  Arms: Face-to-face Group
Other: Control Group — Each of the women will be informed about the purpose and content of the study at the first meeting, and informed consent will be obtained from the women who meet the conditions for participation and agree to participate. The pre-test data in the research will be obtained with the Participant Identification Form and WHOQOL-BREF-TR No intervention will be applied to the mothers in the control group. The end of the 2nd and 6th months, the final test data will be obtained by completing the Participant Identification Form and WHOQOL-BREF-TR
  Arms: Control

SUMMARY:
Introduction: The postpartum period is very important and is a suitable period for women to gain healthy lifestyle behaviors. Studies in the literature show that women with high quality of life have a more comfortable postpartum period. If the needs of women are not met in the postpartum period, there may be an increase in traditional practices for mothers. For this reason, postpartum education is very important for maternal health. Various ways can be used to provide education to mothers. With the development of technology, education given over mobile applications has often found a place in studies. The face-to-face education format, on the other hand, remains up-to-date. It is not known for certain which form of education is superior to the other. Testing the superiority of these two training methods to each other will eliminate the question marks in this area.

Purpose: To determine the effectiveness of WhatsApp-based and face-to-face nursing education and counseling given in the postpartum period on mothers' quality of life and traditional practices.

Method: The experimentally planned study will consist of three groups including WhatsApp, face-to-face and control group. The universe of the research will be composed of women hospitalized in Sivas Numune Hospital Aseptic Service. A total of 180 people will be taken into the sample of the research, 60 of which are in the WhatsApp experimental group, 60 in the face-to-face experimental group and 60 in the control group. Training videos for the postpartum period will be sent to the WhatsApp experimental group via WhatsApp. Face-to-face training will be given to the women in the face-to-face experimental group by the researcher, and the handbook containing the training content will be distributed to the women. Women in both experimental groups will be supported by providing counseling over the phone (message, meeting if needed). No attempt will be made to the control group. The participant introduction form and the Turkish version of the world health organization quality of life scale (WHOQOL-BREF-TR) will be used to evaluate the data of the study. The data will be evaluated with the SPSS 28 program.

DETAILED DESCRIPTION:
After the preliminary test is applied to the experimental groups, Training videos regarding the postpartum period will be sent to the WhatsApp experimental group by the researcher via WhatsApp. Face-to-face training will be given to the women in the face-to-face experimental group by the researcher, and the handbook containing the training content will be distributed to the women. Women in both experimental groups will be supported by providing counseling over the phone (message, meeting if needed).

In the study, training modules including general information about the postpartum period, breastfeeding counseling, postpartum nutrition, puerperal psychology, family planning and postpartum exercises, consisting of 4 sessions, will be applied to the women in the experimental groups. Training module I will be administered within 1 week postpartum; general information about the postpartum period by using the literature (ambulation, hygiene, shower, sexual intercourse time, etc.) and the breastfeeding counseling training that the researcher received from the Ministry of Health (importance of breast milk and breastfeeding, practices that support breastfeeding, the importance of skin-to-skin contact (kangaroo care) etc.) breastfeeding counseling will be given. In the 2nd week, telephone counseling (message, meeting if needed) will be provided and general information about postpartum and possible questions and problems regarding breastfeeding counseling will be evaluated. II. the training module will be implemented at the 3rd postpartum week; By making use of the literature, training and nutrition education (for increasing milk and healthy nutrition, etc.) will be given for postpartum puerperal psychology (postpartum depression, etc.). In the 4th week, possible questions and problems related to the trainings given in the previous weeks will be evaluated by providing counseling by phone (message, interview if needed). III. the training module will be implemented at week 5 postpartum; training on family planning (traditional and modern methods) will be provided by making use of the literature. In the 6th week, possible questions and problems related to the trainings given in the previous weeks will be evaluated by providing counseling by phone (message, interview if needed). IV. and the last training module will be administered at 7 weeks postpartum; By making use of the literature, training on postpartum exercises (aerobics, muscle strengthening, etc.) will be given. In the 8th week, telephone counseling (message, interview if needed) will be provided and possible questions and problems related to the trainings given in the previous weeks will be evaluated. The training contents will be organized according to the health promotion model and expert opinion will be sought regarding the training contents. The trainings will be given to the women in the experimental group face-to-face by the researchers in the form of 15-30 minutes of training in their own home environment.Trainings will be sent to the women in the WhatsApp experimental group in the form of videos via the WhatsApp application. The videos will be prepared with the researchers' own voice and image. Each training video will be sent for 15-30 minutes (in the form of short videos, if necessary, divided into parts).Both experimental groups will be supported through messages to increase the motivation of women and to provide counseling for possible questions and problems.

No intervention will be applied to the mothers in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Be within the first 1 week of the postpartum period,
* Having had a vaginal birth,
* Having a smart phone
* Not having a chronic or psychiatric illness,
* Having given birth at term
* There is no problem with the baby.

Exclusion Criteria:

* Having had a cesarean delivery,
* Not having a smart phone,
* Having a chronic or psychiatric illness,
* Not having given birth at term,
* There is problem with the baby.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
The effect of education given via WhatsApp on traditional postpartum practices | 6 months
  In the first 15 questions of the form, there are questions about the socio-demographic characteristics and obstetric characteristics of the mothers, while the last 9 questions include questions about the traditional methods applied by the mothers.
  In the research, all questions in the participant introduction form and pre-test data will be collected. After completing the scale, mothers will be informed for 2 months, 4 times training and 4 times counseling for 8 weeks. Trainings will be sent from the WhatsApp application and counseling will be provided by phone (message, speaking if necessary). At the end of the 2nd and 6th months, the last 9 questions of the participant introduction form for traditional practices will be asked again.
The effect of education given via WhatsApp on postpartum quality of life | 6 months
  World Health Organization Quality of Life Scale Short Form Turkish Version: The scale consists of 27 questions. High scores from the scale indicate a high quality of life.
  In the research, the pre-test data will be filled with the quality of life scale. After completing the scale, mothers will be informed for 2 months, 4 times training and 4 times counseling for 8 weeks. Trainings will be sent from the WhatsApp application and counseling will be provided by phone (message, speaking if necessary). At the end of the 2nd and 6th months, the quality of life scale will be filled again.
The effect of face-to-face education on traditional postpartum practices | 6 months
  Participant introduction form: In the first 15 questions of the form, there are questions about the socio-demographic characteristics and obstetric characteristics of the mothers, while the last 9 questions include questions about the traditional methods applied by the mothers.
  In the research, all questions in the participant introduction form and pre-test data will be collected. After completing the scale, mothers will be informed for 2 months, 4 times training and 4 times counseling for 8 weeks. The trainings will be given face to face with home visits and consultation will be provided by telephone (message, speaking if necessary). At the end of the 2nd and 6th months, the last 9 questions of the participant introduction form for traditional practices will be asked again.
The effect of face-to-face education on postpartum quality of life | 6 months
  World Health Organization Quality of Life Scale Short Form Turkish Version: The scale consists of 27 questions. High scores from the scale indicate a high quality of life.
  In the research, the pre-test data will be filled with the quality of life scale. After completing the scale, mothers will be informed for 2 months, 4 times training and 4 times counseling for 8 weeks. The trainings will be given face to face with home visits and counseling will be provided by phone (message, speaking if necessary). At the end of the 2nd and 6th months, the quality of life scale will be filled again.

CONTACTS AND LOCATIONS:
Overall Officials: GAMZE DERMAN, Principal Investigator — Inonu University; SERMİN TİMUR TAŞHAN, Professor, Study Director — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No